CLINICAL TRIAL: NCT03160196
Title: Efficacy of an Electronic System to Support Clinical Decisions Based on an Evidence-based Clinical Practice Guide for Metabolic Control of Adults With Type 2 Diabetes Mellitus: Clinical and Cluster-randomized Controlled Trial.
Brief Title: Efficacy of an Electronic System to Support Clinical Decisions in Adults With Type 2 Diabetes Mellitus.
Acronym: OSI-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sanitas University (Other)
Responsible Party: Principal Investigator, Abel Ernesto González Vélez, Principal Investigator, Sanitas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Hemoglobin A, Glycosylated
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental practices (Experimental): The decision support tool is a Web-based software program accessed via a GP computer desktop icon. Clicking the icon opens a single page of tick boxes asking for relevant aspects of the presenting illness. Most fields for relevant medical history and patient demographics are automatically populated from data in the electronic health record. Depending on diagnosis and risk estimation, the tool recommends a guideline-based management strategy. Override options exist but require a justification from the GP. The tool also provides relevant prescriptions, radiology access, and referral forms, and a variety of patient information leaflets. GPs in practices randomized to the intervention group will have to initiate the tool but will not have to follow the tool's advice.
  Interventions: Other: Clinical Decision Support System
- Control practices (Active Comparator): Control practices will be aware of the tool but will be unable to access it and managed patients by usual care, which could include care aligned with the Guidelines. Prior to randomization, GPs from all participating practices (control and intervention) will attend a 1-hour face-to-face didactic education session on diabetes mellitus 2 management and the Colombia diabetes mellitus 2 Guidelines. The intervention pertains to the cluster level.
  Interventions: Other: Usual care based on clinical practice guideline

INTERVENTIONS:
Other: Clinical Decision Support System — It is about a Clinical Decision Support System based on a diabetes mellitus clinical practice guideline.
  Arms: Experimental practices
Other: Usual care based on clinical practice guideline — It is about usual care aligned with the diabetes guideline.
  Arms: Control practices

SUMMARY:
To assess the efficacy of an electronic system to support clinical decisions based on an evidence-based clinical practice guide for metabolic control of adults with Type 2 Diabetes Mellitus through Clinical and cluster-randomized controlled trial in a Colombian population.

ELIGIBILITY:
Inclusion Criteria:

* No prior exposure to the tool (through development and beta testing)
* Access to an organized diabetes pathway consistent with the Sanitas EPS (Entidad Promotora de Salud) diabetes mellitus 2 guideline.

Exclusion Criteria:

* Terminally ill

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1768 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Proportions of participants with normal Hb1Ac | 6 months and a year of enrollment

IPD SHARING:
Plan to Share IPD: No